CLINICAL TRIAL: NCT00544869
Title: Phase 3 Open-label, Study of OPC-41061 in Subjects With Cardiac-induced Edema (Congestive Heart Failure) - an Investigation of the Safety of Treatment Beyond 7 Days and the Effect of Dose Escalation to 30 mg
Brief Title: A Study of OPC-41061 in Subjects With Cardiac-induced Edema (Congestive Heart Failure)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 156-06-006
Record Dates: First submitted 2007-10-15; First posted 2007-10-16 (Estimated); Results first posted 2014-01-30 (Estimated); Last update posted 2014-01-30 (Estimated); Status verified 2013-12

CONDITIONS: Cardiac Edema
Keywords: Vasopressin antagonist , Cardiac Edema ,Diuretics
MeSH Terms: conditions — Edema, Cardiac | interventions — Tolvaptan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: OPC-41061 （Tolvaptan)

INTERVENTIONS:
Drug: OPC-41061 （Tolvaptan) — 15-30mg/day,daily for 14days

SUMMARY:
To investigate the plasma drug level, efficacy, and safety of 7-day repeated oral administration of OPC-41061 at 15 mg/day (treatment period 1) and subsequent 7-day repeated administration of OPC-41061 at 15 mg/day or 30 mg/day if diuretic effect is insufficient (treatment period 2) in congestive heart failure (CHF) patients with extracellular volume expansion despite conventional diuretic therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with cardiac edema receiving diuretic treatment since 7 days prior to the commencement of study drug administration.
2. Subjects receiving one of the following diuretic treatments since 3 days prior to the commencement of study drug administration without changing the dose or dosing regimen (including subjects scheduled to start treatment during the run-in observation period).

   * 1. A loop diuretic at a daily dosage equivalent to 40 mg or more of furosemide
   * 2. Concomitant administration of a loop diuretic and a thiazide diuretic (at any doses)
   * 3. Concomitant administration of a loop diuretic and an anti-aldosterone drug (at any doses)
3. CHF patients with lower limb edema, jugular venous distention, or pulmonary congestion due to extracellular volume expansion.
4. Male or female subjects between the ages of 20 and 85, inclusive (at time of informed consent)
5. Subjects able to stay at the study site from the day before the start of the run-in observation period until completion of post-treatment observation 2 (7 to 10 days after final study drug administration)
6. Subjects capable of giving informed consent to participate in the study of their own free will

Exclusion Criteria:

1. Heart failure patients with markedly fluctuating symptoms
2. Patients with an assisted circulation device
3. Patients with any of the following complications or symptoms:

   * 1. Suspected decrease in circulatory blood flow ，
   * 2. Hypertrophic cardiomyopathy (other than dilated phase)，
   * 3. Cardiac valve disease with significant heart valve stenosis，
   * 4. Hepatic coma
4. Patients who develop acute myocardial infarction within 30 days prior to the screening examination
5. Patients with a definite diagnosis of active myocarditis or amyloid cardiomyopathy
6. Subjects with any of the following complications or symptoms:

   * 1. Poorly controlled diabetes melllitus，
   * 2. Anuria，
   * 3. Urination impaired due to urinary tract stricture, urinary calculus, tumor in urinary tract, or other cause
7. Subjects with any of the following disease histories:

   * 1. Sustained ventricular tachycardia or ventricular fibrillation within 30 days prior to the screening examination in subjects without an implanted defibrillator，
   * 2. Cerebrovascular disorder within 6 months prior to the screening examination (other than asymptomatic cerebral infarction)，
   * 3. A history of hypersensitivity or idiosyncratic reaction to benzazepine derivatives such as mozavaptan hydrochloride or benazepril hydrochloride.
8. Subjects who are severely obese [body mass index (BMI, body weight (kg)/height (m)2] exceeding 35]
9. Subjects with systolic blood pressure in the decubitus position exceeding 90 mmHg
10. Subjects with any of the following abnormal laboratory values:

    * 1. Total bilirubin > 3.0 mg/dL,
    * 2. serum creatinine > 3.0 mg/dL,
    * 3. serum sodium > 147 mEq/L,
    * 4. serum potassium > 5.5 mEq/L
11. Patients who are unable to take oral medication
12. Female subjects who are pregnant, possibly pregnant, or lactating, or who plan to become pregnant during the study period
13. Subjects who received any investigational drug other than OPC-41061 within 30 days prior to the screening examination
14. Subjects otherwise judged by the investigator or subinvestigator to be inappropriate for inclusion in the study

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2007-10; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katsuhisa Saito, Study Director — Division of New Product Evaluation and Development
Locations (6):
- Japan (6):
  - Chubu Region
  - Hokkaido Region
  - Kanto Region
  - Kinki Region
  - Kyuush
  - Shikoku Region

RESULTS

PARTICIPANT FLOW:
Groups:
- Stopped at End of Treatment Period 1: Administration of OPC-41061 at 15 mg/day (treatment period 1) for 7 days
- Continued at 15 mg/Day: Subsequent 7-day repeated administration of OPC-41061 at 15 mg/day (treatment period 2)
- Dose Escalated to 30 mg/Day: Subsequent 7-day repeated administration of OPC-41061 at 30 mg/day (treatment period 2)
Period: Overall Study
Arm/Group | Stopped at End of Treatment Period 1 | Continued at 15 mg/Day | Dose Escalated to 30 mg/Day
Started | 36 | 14 | 2
Completed | 24 | 12 | 2
Not Completed | 12 | 2 | 0
Not completed — Rsolution of congenitive symptoms | 3 | 0 | 0
Not completed — Adverse Event | 6 | 1 | 0
Not completed — Lack of Efficacy | 1 | 1 | 0
Not completed — Physician Decision | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: 1 Subject of Arm "Continued at 15 mg/day" was excluded from analysis because of GCP incompliance
Groups:
- Total: Total of all reporting groups
Arm/Group | Stopped at End of Treatment Period 1 | Continued at 15 mg/Day | Dose Escalated to 30 mg/Day | Total
Number analyzed (Participants) | 36 | 13 | 2 | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 4 | 0 | 11
  >=65 years | 29 | 9 | 2 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.3 (9.5) | 67.2 (12.7) | 78.5 (2.1) | 70.5 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 2 | 1 | 14
  Male | 25 | 11 | 1 | 37
Region of Enrollment [Number; unit: participants]
  Japan | 36 | 13 | 2 | 51

OUTCOME MEASURES:

1. Primary Outcome: Body Weight
Description: The change of body weight from baseline at final observation
Time Frame: Baseline, Day 14 or at the time of final drug administration
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | Stopped at End of Treatment Period 1 | Continued at 15 mg/Day | Dose Escalated to 30 mg/Day
Number analyzed (Participants) | 36 | 13 | 2
Kg | -2.05 (1.86) | -1.31 (2.95) | -2.9 (2.69)

ADVERSE EVENTS:
Time Frame: 7 Days for stopped at end of treated period 1 group 14 Days for continued at 15 or 30 mg/day group
Arm/Group | Stopped at End of Treatment Period 1 | Continued at 15 mg/Day | Dose Escalated to 30 mg/Day
Serious Adverse Events (participants affected / at risk) | 3/36 | 1/13 | 0/2
Other Adverse Events (participants affected / at risk) | 30/36 | 12/13 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stopped at End of Treatment Period 1 (N=36) | Continued at 15 mg/Day (N=13) | Dose Escalated to 30 mg/Day (N=2)
Cardiac Failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Intracardiac Thrombus (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebral Artery Embolism (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Renal Failure Chronic (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stopped at End of Treatment Period 1 (N=36) | Continued at 15 mg/Day (N=13) | Dose Escalated to 30 mg/Day (N=2)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac Failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Ventricular Extrasystoles (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Ventricular Tachycardia (Cardiac disorders) | 4 (4) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 1 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 5 (5) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
Chest Pain (General disorders) | 2 (2) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Thirst (General disorders) | 14 (14) | 6 (6) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Alanine Aminotransferase Increased (Investigations) | 3 (3) | 0 (0) | 0 (0)
Aspartate Aminotransferase Increased (Investigations) | 3 (3) | 1 (1) | 0 (0)
Blood Alkaline Phosphatase Increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood Creatinine Increased (Investigations) | 4 (4) | 4 (4) | 1 (1)
Blood Glucose Increased (Investigations) | 4 (4) | 4 (4) | 0 (0)
Blood Lactate Dehydrogenase Increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood Potassium Increased (Investigations) | 3 (3) | 3 (3) | 0 (0)
Blood Urea Increased (Investigations) | 6 (6) | 4 (4) | 1 (1)
Blood Uric Acid Increased (Investigations) | 6 (6) | 4 (5) | 1 (1)
Blood Urine Present (Investigations) | 1 (1) | 1 (1) | 0 (0)
Glucose Urine Present (Investigations) | 1 (1) | 1 (1) | 0 (0)
White Blood Cell Count Increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0)
Renal Impairment (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 0 (0)
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Haemorrhage Subcutaneous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No